CLINICAL TRIAL: NCT02556658
Title: Predicted Level of General Anaesthesia in Hip Fracture Surgery
Acronym: NAPfem
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2014-A01243-44
Record Dates: First submitted 2015-01-21; First posted 2015-09-22 (Estimated); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Hip Fracture Surgery
Keywords: Smartpilot View; Hip fracture surgery; Depth of anaesthesia; Intraoperative hypotension; Quality of anaesthesia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Smartpilot View group (Experimental): General anaesthesia managed by the Smartpilot® View device The intervention consists of administering hypnotics and opioids according to effect-site concentrations and interaction model provided by the Smartpilot® View software for the entire duration of general anaesthesia.
  Interventions: Device: General anesthesia managed by the Smartpilot® View
- Control group (Active Comparator): General anaesthesia without using the Smartpilot® View device The anesthetic induction will be performed by propofol or sufentanil and atracurium. The maintenance of anesthesia will be directed by desflurane and sufentanil. The dosages of anesthetics are left to the discretion of the doctor and nurse anesthetists in charge of the patient in the operating room.
  Interventions: Device: General anesthesia managed without the Smartpilot® View

INTERVENTIONS:
Device: General anesthesia managed by the Smartpilot® View — General anaesthesia managed by the Smartpilot® View device The intervention consists of administering hypnotics and opioids according to effect-site concentrations and interaction model provided by the Smartpilot® View software for the entire duration of general anaesthesia.
  Arms: Smartpilot View group
Device: General anesthesia managed without the Smartpilot® View — General anaesthesia without using the Smartpilot® View device The anesthetic induction will be performed by propofol or sufentanil and atracurium. The maintenance of anesthesia will be directed by desflurane and sufentanil. The dosages of anesthetics are left to the discretion of the doctor and nurse anesthetists in charge of the patient in the operating room.
  Arms: Control group

SUMMARY:
The purpose of this study is to evaluate if prediction of general anaesthesia level by the Smartpilot® View device can improve the quality of anaesthesia in patients undergoing hip fracture surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing hip fracture surgery under general anaesthesia
* Age ≥ 18 years old
* ASA classification 1, 2 or 3

Exclusion Criteria:

* Patient not insured by a social security scheme
* Adult patient under tutorship or curatorship
* Age over 18 years old or under 90 years old
* Weight under 40 or over 140 kilos and/or height under 150 or over 200 cm
* Body mass index > 35
* Contraindication to one or more anaesthetics used in the study
* Pregnancy or breastfeeding
* Unweaned alcoholism
* ASA classification 4 or 5
* Patient undergoing hip fracture surgery under spinal anaesthesia

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-02; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Percentage of time spent in the "appropriate anaesthesia zone" | participants will be followed for the duration anesthesia, an expected average of 5 hours (from intubation to recovery) for hip fracture surgery
  The "appropriate anaesthesia zone" is defined as a bispectral index between 45 and 65 and a systolic blood pressure between 80 and 140 mmHg

SECONDARY OUTCOMES:
Dose of propofol | participants will be followed for the duration anesthesia, an expected average of 5 hours
Dose of sufentanil | participants will be followed for the duration anesthesia, an expected average of 5 hours
Time to extubation | end of anaesthesia
"NASA Task Load Index" | participants will be followed for the duration anesthesia, an expected average of 5 hours
Morphine consumption | participants will be followed for the duration in recovery room, an expected average of 24 hours
Incidence of awareness with recall during anaesthesia | postoperative day 1
"Postoperative Quality Recovery Scale" | during recovery room (an expected average of 24 hours) and postoperative days 1 and 3
Length of stay | postoperative day 30
Mortality | postoperative day 30

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu CONTE, M.D., Principal Investigator — University Hospital, Angers
Locations (1):
- University Hospital Angers, Angers, France

REFERENCES:
- [Result] Leblanc D, Conte M, Masson G, Richard F, Jeanneteau A, Bouhours G, Chretien JM, Rony L, Rineau E, Lasocki S. SmartPilot(R) view-guided anaesthesia improves postoperative outcomes in hip fracture surgery: a randomized blinded controlled study. Br J Anaesth. 2017 Nov 1;119(5):1022-1029. doi: 10.1093/bja/aex317. PMID 29028921